CLINICAL TRIAL: NCT00577746
Title: The Clinical Impact of Endoscopic Ultrasound (EUS) in Staging Non-small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Impact of EUS in Staging NSCLC
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Richard L. Roudebush VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0306-37; IRB # 0306-37
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung
Keywords: Non Small Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- surgery: Those subjects who went to surgery for treatment for their lung cancer.
- no surgery: The subjects who did not go to surgery for treatment of their lung cancer.

SUMMARY:
The goal of this prospective study is to determine the clinical and economic impact of endoscopic ultrasound (EUS) in staging NSCLC. Aims: 1) Determine the accuracy of EUS in staging NSCLC 2) Measure 5-year survival 3) Measure quality of life in patients that undergo surgery 4) Determine the cost benefit of EUS in staging NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with presumed or known potentially resectable NSCLC
* Due to the nature of NSCLC, children (<18 year of age) will not be considered
* Men, women, and minorities
* Subjects must be able to safely undergo conscious sedation for the EUS procedure
* Subjects must be surgical candidates
* Subjects must not have an uncorrectable coagulopathy and must be able to refrain from the used of aspirin one week prior to the EUS
* Patient must provide signed written informed consent

Exclusion Criteria:

* Subjects with a history of previously treated lung, head & neck, or esophageal cancer are not eligible if the histologic cell type is determined to be the same as what is biopsied during the EUS-FNA
* Uncorrectable coagulopathy
* Significant co-morbidities such as uncontrolled heart failure, or severe chronic obstructive pulmonary disease (COPD) that would limit their survivability to surgery
* Evidence of significant active infection (e.g. pneumonia, peritonitis, wound abscess)
* Evidence of serious ongoing illness such as uncontrolled metabolic disease (diabetes mellitus, hypothyroidism, etc.) or cardiac condition
* Evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric illness that would preclude adequate compliance with this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially resectable lung cancer subjects see at thoracic oncology clinics and gastroenterolgy lab.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2006-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determine the accuracy of EUS in staging NSCLC | at the end of the study

SECONDARY OUTCOMES:
Measure 5-year survival | 5 years
Determine the cost benefit of EUS in staging NSCLC | at the end of the study
Measure quality of life in patients that undergo surgery | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Medical Center; Clarian Health, Indianapolis, Indiana, United States